CLINICAL TRIAL: NCT05771948
Title: Effectiveness and Safety of CCoat Intra-Articular Injections in Mild to Moderate Knee Osteoarthritis: Prospective, Placebo Controlled, Randomized, Double-Blinded Study
Brief Title: Effectiveness and Safety of CCoat Intra-Articular Injections in Mild to Moderate Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lipo-Sphere (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLD-0000616
Record Dates: First submitted 2023-03-05; First posted 2023-03-16 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Control) (Placebo Comparator): 1 IA injection of 4 ml Normal Saline solution.
  Interventions: Device: CCoat
- Group 2 (Study) (Experimental): 1 IA injection of 4 ml CCoat
  Interventions: Device: CCoat

INTERVENTIONS:
Device: CCoat — CCoat is a new intra-articular (IA) injectable joint lubricant for patients suffering from joint pain developed by Liposphere LTD. CCoat is a liposomal boundary lubricant which coats the cartilage surface and protects it from further damage and degradation.

SUMMARY:
The goal of this clinical trial is to evaluate the Efficacy and Safety of CCoat Intra-Articular Injection in Mild to Moderate Knee Osteoarthritis.

The main questions it aims to answer are:

* To demonstrate superior efficacy of CCoat administered via intra-articular injection versus placebo during the study period.
* To evaluate the efficacy of two different concentrations of CCoat, administered via single IA injection as compared to control group (placebo) One IA injection of CCoat or Placebo will be injected to participants' knee. Follow up will take place up to six months.
* To evaluate the safety of the repeated CCoat injection administered at six months.

DETAILED DESCRIPTION:
This study aims to assess the effectiveness and safety of intra-articular injection of Aqueous Joint at two different concentrations administered via a single injection in osteoarthritic patients up to 26 weeks of follow-up in a double-blind, randomized clinical study. Additionally, the safety of the repeated injection will be examined.

Primary Effectiveness Objective The primary objective is to demonstrate the superior effectiveness of CCoat administered via single intra-articular injection versus placebo during the study period in terms of functional outcomes as assessed in terms of Pain KOOS subscore at each FU visit (up to and including 12 weeks) and compared to the baseline levels.

Secondary Effectiveness Objective The secondary objective is to assess changes from baseline to 26 weeks in NRS, KOOS symptoms, QOL, ADL and sport subscores. Change from Baseline in Patient's Global Assessment (PGA)) of Osteoarthritis at Week 26 were evaluated. Patients responder rates will be evaluated at 12 and 26 weeks.

Safety Objectives Safety will be evaluated by the occurrence of Adverse Events during the study. Adverse Events will be reported in terms of incidence, severity, and frequency of all Adverse Events (AE).

Clinical Hypotheses The underlying clinical hypothesis of this study is that the CCoat is superior to the control group in terms of KOOS score (Pain, Symptoms, QOL, ADL & Sports) at 3 months compared to baseline, even more in a high concentration.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated the informed consent form
2. Age ≥30 and ≤ 85 years old
3. Pain in the intended study knee with an average VAS score (active) of ≥3 over the last week before screening.
4. Degenerative changes in the intended study knee that can be categorized as grade I -III- Kellgren Lawrence based upon standing anterior- posterior and lateral radiographsof the knee
5. Body Mass Index (BMI) between 18.5 and 38
6. A negative urine pregnancy test female patient with childbearing potential at Visit 1 prior to intra-articular injection of AqueousJoint.
7. If female, the subject must be either postmenopausal, OR permanently surgically sterile OR for women of childbearing potential using at least 2 methods of birth control that are effective from at least 30 days before Visit 1 through visit 26w (26 weeks post injection).
8. Are willing or able to comply with procedures required in this protocol.

Exclusion Criteria:

1. Osteoarthritis of the index knee graded 4 according to the Kellgren-Lawrence Grading
2. History of significant knee trauma or previous surgery of the intended study knee within the last 3 months preceding the screening
3. Pain in both knees with a VAS score of ≥5
4. Intra-articular injection to the intended study knee within 3 months before Screening
5. Significant instability of the index knee
6. Malalignment more than 10 degrees varus OR 10 degrees valgus according to standing X-ray
7. Intake of chronic pain medications (especially opioid pain relievers) without an option to pause for the period of the study
8. History of Psoriatic Arthritis, Rheumatoid Arthritis, or any other inflammatory condition associated with arthritis
9. Wound in the area of the intended study knee
10. Any known tumor of the index knee
11. Any known history of intra-articular or osseous infection of the index knee
12. Any evidence of active infection anywhere in the body. Urinary Tract Infection (UTI) patients can be included following antibiotic treatment, provided that two consecutive cultures are negative (taken within at least 2 weeks of each other)
13. Any known history of inflammatory arthropathy or crystal-deposition arthropathy
14. Any known systemic cartilage and/or bone disorder, such as but not limited to, chondrodysplasia or osteogenesis imperfecta
15. Body Mass Index (BMI) > 38
16. Active malignances, excluding BCC.
17. Chemotherapy and/or radiation in the past 12 months
18. Known history of a severe allergic reaction
19. Patient who is pregnant or intends to become pregnant during the study
20. History of any significant systemic disease, such as but not limited to: HIV, hepatitis, HTLV, syphilis, and coagulopathies
21. A Known substance or alcohol abuse
22. Participation in other clinical trials within 60 days to before the study or concurrent with the study
23. Known insulin dependent diabetes mellitus
24. Unable to undergo X-ray

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) PAIN | Baseline up to 12 weeks
  Change from baseline in patients KOOS pain over the course of the 12-week initial treatment period as measured by using the Knee injury and Osteoarthritis Outcome Score (KOOS) in following subscore: Pain- [Time Frame: Day 0, up to week 12]
  The responses for the KOOS Pain subscale are then summed and transformed into a score ranging from 0 to 100, where:
  0 represents extreme problems (maximum pain) 100 represents no problems (no pain)

SECONDARY OUTCOMES:
Numerical Rating Scale (NRS) Pain Score | Assessed at1, 6, 12, and 26 weeks from baseline.
  Change in Numerical Rating Scale (NRS) Pain.
  The NRS asks patients to rate their pain on a scale from 0 to 10, where:
  0 represents "No pain" 10 represents "Worst possible pain"
PGA | Baseline to 6,12 and26 weeks
  Change in Patient's Global Assessment (PGA). PGA assessment includes 5 options to answer - between 1 to 5 - which 1 means 'very good' , and 5 means 'very poor'.
Knee Injury and Osteoarthritis Outcome Score Responder Rates | Baseline to 12 weeks
  A responder is defined as an improvement of at least 8 points or ≥ 20% from baseline in the each of the KOOS subscores (Pain; Activities of Daily Living (ADL);Quality of Life (QOL);Symptoms; Sports; Overall KOOS score)
  The MCID is the smallest change in a score that patients perceive as beneficial. For the KOOS, an improvement of around 8 points in a subscale score is often considered a clinically meaningful change.
  A patient might be considered a responder if they achieve at least the MCID in one or more of the KOOS subscales (Pain, ADL, Sports, Symptoms, QOL).
Subscores-Specific KOOS Improvements | Baseline to 6,12 and26 weeks
  Measured Change in the following KOOS subscores ( pain, ADL, sports, symptoms, QOL)
  Each of the five KOOS subscales is scored separately on a scale from 0 to 100, where 0 represents extreme problems and 100 represents no problems.
  Calculate the Change:
  Subtract the baseline score from the follow-up score for each subscale. Change in KOOS Subscale = Follow-Up Score - Baseline Score A positive change indicates improvement (e.g., less pain, better ADL, better sports function).
  A negative change indicates worsening (e.g., more pain, worse ADL).
Safety | baseline to 6 month
  Adverse events, including serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Michael Drexler, Prof., Principal Investigator — Orthopedic department
Locations (3):
- Israel (3):
  - Assuta, Ashdod
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot

IPD SHARING:
Plan to Share IPD: No